CLINICAL TRIAL: NCT02086006
Title: A NON-RANDOMIZED, CONSECUTIVE ENROLLMENT EVALUATION OF THE DESolveTM MYOLIMUS ELUTING BIORESORBABLE CORONARY STENT SYSTEM IN THE TREATMENT OF PATIENTS WITH DE NOVO NATIVE CORONARY ARTERY LESIONS
Brief Title: Elixir Medical Clinical Evaluation of the DESolve Myolimus Eluting Bioresorbable Coronary Stent System - DESolve I Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1002
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DESolve scaffold (Other): DESolve Novolimus Eluting Bioresorbable Coronary Scaffold. test arm, intervention
  Interventions: Device: DESolve Novolimus Eluting Bioresorbable Coronary Scaffold

INTERVENTIONS:
Device: DESolve Novolimus Eluting Bioresorbable Coronary Scaffold

SUMMARY:
This prospective, consecutive enrolment, single-arm study will enroll up to 15 patients with single de novo, Type A lesions < 10 mm in length and located in a native coronary artery with a reference vessel diameter of 2.75 mm - 3.0 mm as measured by both offline QCA and IVUS. All patients will receive a 3.0 x 14mm DESolve Stent loaded with approximately 40 mcg of Myolimus.

* Angiographic and intravascular ultrasound (IVUS) will be completed for all patients at baseline and at 6 months.
* Optical Coherence Tomography (OCT) will will be completed for all patients at baseline and at 6 months.
* Multi-slice computed tomography (MSCT) will be conducted on all patients enrolled at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the DESolve Myolimus Eluting BCSS and he/she or his/her legally authorized representative provides written informed consent, as approved by the appropriate Ethics Committee of the respective clinical site, prior to any clinical study related procedure
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study electrocardiogram (ECG) changes consistent with ischemia)
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery
* Patient must agree to undergo all clinical study required follow-up visits, angiograms, IVUS, OCT and MSCT
* Patient must agree not to participate in any other clinical study for a period of two years following the index procedure

Exclusion Criteria:

* Patients has a known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure and CK and CK-MB have not returned within normal limits at the time of procedure
* The patient is currently experiencing clinical symptoms consistent with AMI
* Patient has current unstable arrhythmias Patient has undergone previous percutaneous interventions for lesions in either a non-target vessel or target vessel Patient has undergone previous percutaneous interventions for lesions in either a non-target vessel or target vessel
* Patient has a known left ventricular ejection fraction (LVEF) < 30%
* Patient has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant
* Patient is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or after the procedure
* Patient is receiving immunosuppression therapy and has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.)
* Patient is receiving or scheduled to receive chronic anticoagulation therapy (e.g., heparin, coumadin)
* Patient has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, both clopidogrel and ticlopidine, Myolimus, PLLA polymers or contrast sensitivity that cannot be adequately pre-medicated
* Elective surgery is planned within the first 6 months after the procedure that will require discontinuing either aspirin or clopidogrel
* Patient has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3, or documented or suspected liver disease.
* Patient has known renal insufficiency (e.g., serum creatinine level of more than 2.5 mg/dL, or patient on dialysis)
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic neurological attack (TIA) within the past six months
* Patient has had a significant GI or urinary bleed within the past six months
* Patient has extensive peripheral vascular disease that precludes safe 7 French sheath insertion
* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical study plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
* Patient is already participating in another clinical study
* Women of childbearing potential who have not undergone surgical sterilization or is not post-menopausal (defined as amenorrheic for at least one year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 1 month
Clinically-Indicated Target Lesion Failure (CI-TLF) | 1 month
Clinically-Indicated Target Vessel Failure (CI-TVF) | 1 month
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 1 month
Stent thrombosis | 1 month
Acute success - Procedure success | 7 days
  Acute Success is classified according to the following definitions:
  Procedure success - Attainment of final result, < 50% residual stenosis of the target site, using the DESolve Myolimus Eluting BCSS device without the occurrence of in-hospital any Major Adverse Cardiac Endpoints.
Acute success - Device success | 7 days
  Acute Success is classified according to the following definitions:
  Device success - Attainment of final result, < 50% residual stenosis of the target site, using the study stent without the need for other non-study stents.
Stent thrombosis | 6 months
Stent thrombosis | 12 months
Stent thrombosis | 2 years
Stent thrombosis | 3 years
Stent thrombosis | 4 years
Stent thrombosis | 5 years
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 6 months
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 12 months
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 2 years
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 3 years
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 4 years
Clinically-Indicated Major Adverse Cardiac Event (CI-MACE) | 5 years
Clinically-Indicated Target Lesion Failure (CI-TLF) | 6 months
Clinically-Indicated Target Lesion Failure (CI-TLF) | 12 months
Clinically-Indicated Target Lesion Failure (CI-TLF) | 2 years
Clinically-Indicated Target Lesion Failure (CI-TLF) | 3 years
Clinically-Indicated Target Lesion Failure (CI-TLF) | 4 years
Clinically-Indicated Target Lesion Failure (CI-TLF) | 5 years
Clinically-Indicated Target Vessel Failure (CI-TVF) | 6 months
Clinically-Indicated Target Vessel Failure (CI-TVF) | 12 months
Clinically-Indicated Target Vessel Failure (CI-TVF) | 2 years
Clinically-Indicated Target Vessel Failure (CI-TVF) | 3 years
Clinically-Indicated Target Vessel Failure (CI-TVF) | 4 years
Clinically-Indicated Target Vessel Failure (CI-TVF) | 5 years
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 6 months
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 12 months
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 2 years
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 3 years
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 4 years
Clinically-Indicated Target Vessel Revascularization (CI-TVR) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Ormiston, MD, Principal Investigator — Auckland City Hospital and Mercy Angiography Unit; Stefan Verheye, MD, PhD, Principal Investigator — ZNA Middelheim
Locations (3):
- AZ Middelheim Hospital, Antwerp, Belgium
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Mercy Angiography Unit, Auckland